CLINICAL TRIAL: NCT01990144
Title: Rituximab Plus Bendamustine as Front Line Treatment in Frail Elderly (>70 Years) Patients With Diffuse Large B-cell Non-Hodgkin's Lymphoma: a Phase II Multicenter Study of the Fondazione Italiana Linfomi (FIL)
Brief Title: Rituximab Plus Bendamustine as Front Line Treatment in Frail Elderly (>70 Years) Patients With DLBCL: a Phase II Multicenter Study of the FIL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_R-BENDA FRAIL
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bendamustine (Experimental): Bendamustine is a novel chemotherapeutic agent, a hybrid of a purine analogue and an alkylator. It shows only partial in vitro cross-resistance with other alkylating agents and it is clinically well tolerated. In fact it has shown to be active in vitro against cell lines which are resistant to other alkylating agents. Preclinical data demonstrate that bendamustine acts in two distinct ways to kill cancer cells: it damages the DNA in cancer cells, which leads to cell death by a process known as apoptosis (programmed cell death) as well as by an alternate cell death pathway known as mitotic catastrophe (a disruption of normal cell division). This dual-effect may be attributable to its unique chemical structure.Bendamustine has demonstrated clinical activity in patients with chronic lymphocytic leukaemia, patients with relapsed indolent NHL, mantle cell lymphoma, multiple myeloma and several solid tumors.
  Interventions: Drug: Bendamustine+Rituximab

INTERVENTIONS:
Drug: Bendamustine+Rituximab — Patients will receive :
  * Rituximab 375 mg/m2 intravenously on day 1*
  * Bendamustine 90 mg/m2 intravenously on days 2 and 3** Treatment will be administered on a 28-day cycle basis.
    * Administration of rituximab during cycle 1 is postponed to day 8, thereafter on day 1.
      * After the first cycle, bendamustine can be administered on days 1-2 or days 2-3 according to Institutional/patient/physician choice.

SUMMARY:
The purpose of the study is to evaluate feasibility and efficacy of rituximab-bendamustine (R-B)combination in elderly patients affected by diffuse large B-cell lymphoma and defined as frail according to CGA.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven CD20 positive diffuse large B-cell non-Hodgkin's lymphoma
* Age > 70 years
* No previous treatment
* FRAIL patients defined as follows (see Appendices B-E) Age > 80 years with UNFIT profile, i.e.

  * ADL > 5 residual functions
  * IADL > 6 residual functions
  * CIRS 5-8 co-morbidities of grade 2

or Age < 80 years with

* ADL < 4 residual functions, or
* IADL < 5 residual functions, or
* CIRS : 1 co-morbidity of grade 3-4, or > 8 co-morbidities of grade 2

  * Life expectancy > 6 months
  * Written informed consent
  * Accessibility of patient for treatment and follow up

Exclusion Criteria:

* History of other malignancies within 5 years prior to study entry except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer
* Previous exposure to cytotoxic agents
* Suspect or clinical evidence of CNS involvement by lymphoma
* HBsAg, HCV or HIV positivity; HBcAb positivity is accepted only with concomitant treatment with Lamivudine
* AST /ALT > twice upper the normal range; bilirubin > twice upper the normal range; serum creatinine > 2.5 mg /dl
* Evidence of any severe active acute or chronic infection
* Concurrent co-morbid medical condition which might exclude administration of full dose chemotherapy
* Senile dementia
* Any other co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the activity of R-B combination in terms of complete response rate (CRR). | 4 years
To evaluate the safety and tolerability of R-B combination in terms of rate of adverse events occurrence. | 4 years

SECONDARY OUTCOMES:
To evaluate progression free survival (PFS) | 4 years
To evaluate overall survival (OS) | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Michele Spina, MD, Principal Investigator — IRCCS CENTRO DI RIFERIMENTO ONCOLOGICO (CRO) - AVIANO (PN)
Locations (52):
- Italy (52):
  - Ospedale Civile Ss. Antonio E Biagio Di Alessandria, Alessandria, Alessandria
  - Ente Eccl.Osp.Gen.Reg.'Miulli', Acquaviva delle Fonti, Bari
  - Ospedale S. Nicola Pellegrino Di Trani, Trani, Barletta
  - Asp Di Bolzano - Comprensorio Sanitario Di Bolzano, Bolzano, Bolzano
  - Pres.Ospedal.Spedali Civili Brescia, Brescia, Brescia
  - Stabilimento "Perrino", Brindisi, Brindisi
  - Ospedale Armando Businco -, Cagliari, Cagliari
  - A.O. Universitaria Ospedale Vittorio Emanuele E Ferrarotto Di Catania, Catania, Catania
  - Nuovo Ospedale Garibaldi - Nesima, Catania, Catania
  - Osp.Generale Di Zona Valduce, Como, Como
  - Presidio Ospedaliero Annunziata, Cosenza, Cosenza
  - Irccs Ospedale Casa Sollievo Della Sofferenza, San Giovanni Rotondo, Foggia
  - Irst - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori, Meldola, Forlì-Cesena
  - A.O. Universitaria S. Martino Di Genova, Genova, Genova
  - Ospedale Generale Di Zona, Civitanova Marche, Macerata
  - Presidio Ospedaliero Matera, Matera, Matera
  - A.O. Universitaria Policlinico Martino Di Messina, Messina, Messina
  - Azienda Ospedaliera Papardo, Messina, Messina
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Milano
  - Ospedale S. Carlo Borromeo, Milan, Milano
  - Ospedale Ca' Granda-Niguarda, Milan, Milano
  - A.O. Universitaria Policlinico Di Modena, Modena, Modena
  - Nuovo Ospedale Di Sassuolo S.P.A., Sassuolo, Modena
  - Azienda Ospedaliera S. Gerardo Di Monza, Monza, Monza
  - Irccs Istituto Oncologico Veneto (Iov), Padua, Padova
  - A.O. Universitaria Policlinico Giaccone Di Palermo, Palermo, Palermo
  - A.O. "V. Cervello", Palermo, Palermo
  - Casa Di Cura La Maddalena Di Palermo, Palermo, Palermo
  - A.O. Universitaria Di Parma, Parma, Parma
  - Ospedale Civile Spirito Santo, Pescara, Pescara
  - Ausl Di Piacenza, Piacenza, Piacenza
  - A.O. Universitaria Pisana, Pisa, Pisa
  - Irccs Centro Di Riferimento Oncologico (Cro), Aviano, Pordenone
  - Irccs Centro Di Riferimento Oncologico Di Basilicata (Crob), Rionero in Vulture, Potenza
  - Ospedale S. Maria Delle Croci Di Di Ravenna, Ravenna, Ravenna
  - Ospedale Bianchi - Melacrino - Morelli, Reggio Calabria, Reggio Calabria
  - Ospedale Di S. Maria Nuova, Reggio Emilia, Reggio Emilia
  - Ospedale Di Rimini, Rimini, Rimini
  - Irccs Istituto Regina Elena (Ifo), Roma, Roma
  - Ospedale S. Eugenio, Roma, Roma
  - Azienda Osp. S.Giovanni/Addolorata Roma, Roma, Roma
  - P.O. Umberto I, Nocera Inferiore, Salerno
  - A.O.Oo.Rr.S.Giovanni Di Dio E Ruggi D'Ar, Salerno, Salerno
  - A.O. Universitaria Policlinico Di Sassari, Sassari, Sassari
  - A.O. Universitaria Senese, Siena, Siena
  - Stabilimento Ss. Annunziata, Taranto, Taranto
  - Azienda Ospedaliera "S. Maria", Terni, Terni
  - Ospedale Civile Di Ivrea, Ivrea, Torino
  - Ematologia 1 - A.O. UNIVERSITARIA S. GIOVANNI BATTISTA-MOLINETTE DI TORINO, Torino, Torino
  - Ematologia 2 - A.O. UNIVERSITARIA S. GIOVANNI BATTISTA-MOLINETTE DI TORINO, Torino, Torino
  - Ematologia - OSPEDALE DI CIRCOLO E FONDAZIONE MACCHI, Varese, Varese
  - Oncologia - OSPEDALE DI CIRCOLO E FONDAZIONE MACCHI, Varese, Varese

REFERENCES:
- [Derived] Storti S, Spina M, Pesce EA, Salvi F, Merli M, Ruffini A, Cabras G, Chiappella A, Angelucci E, Fabbri A, Liberati AM, Tani M, Musuraca G, Molinari A, Petrilli MP, Palladino C, Ciancia R, Ferrario A, Gasbarrino C, Monaco F, Fraticelli V, De Vellis A, Merli F, Luminari S. Rituximab plus bendamustine as front-line treatment in frail elderly (>70 years) patients with diffuse large B-cell non-Hodgkin lymphoma: a phase II multicenter study of the Fondazione Italiana Linfomi. Haematologica. 2018 Aug;103(8):1345-1350. doi: 10.3324/haematol.2017.186569. Epub 2018 May 10. PMID 29748444